CLINICAL TRIAL: NCT00469274
Title: A Randomized Open-Label Non-Inferiority Study to Examine the Impact of Pertussis Vaccination of Healthcare Workers on Post-exposure Prophylaxis
Brief Title: Vanderbilt Pertussis Exposure Study: PEP in Vaccinated Healthcare Workers Following Pertussis Exposure
Acronym: VPES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Tom Talbot, Associate Professor of Medicine, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VPES
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Results first posted 2013-01-29 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2012-12

CONDITIONS: Pertussis
Keywords: Pertussis; Healthcare worker; Post-exposure prophylaxis; Vaccination; Pertussis in healthcare workers following occupational; exposure to pertussis
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antibiotic PEP (Active Comparator): Subjects who did receive PEP following pertussis exposure
  Interventions: Drug: Antibiotic PEP
- No PEP (No Intervention): Subjects who did not receive PEP following pertussis exposure

INTERVENTIONS:
Drug: Antibiotic PEP — Azithromycin 1000mg po x 1, then 500mg po Q day for 4 days; TMP-SMX DS one BID for 14 days
  Arms: Antibiotic PEP
Drug: Antibiotic PEP — TMP-SMX DS po BID for 14 days
  Arms: Antibiotic PEP

SUMMARY:
The purpose of this study is to compare the effectiveness of two strategies of post-exposure prophylaxis (PEP) in healthcare workers (HCWs) who have been vaccinated with acellular pertussis vaccine and have been exposed to pertussis Secondary Objectives include a comparison of the costs of each PEP strategy and an assessment for risk factors associated with healthcare-associated acquisition of pertussis.

DETAILED DESCRIPTION:
Pertussis, caused by the bacterium Bordetella pertussis, is an acute respiratory tract infection transmitted to susceptible persons through aerosolized respiratory droplets and direct contact with respiratory secretions. Classic pertussis disease is characterized by three phases of illness: the catarrhal phase where persons note cough and coryza; the paroxysmal phase where persons develop a spasmodic cough with post-tussive vomiting and an inspiratory whoop; and the convalescent phase, during which symptoms slowly resolve. The risk of transmission of the organism is compounded by the nondescript nature of symptoms early in the course of illness, particularly in adults. Classically recognized as a disease of infants and children ("whooping cough"), the incidence of pertussis infection in adolescents and adults has increased in recent years. Persons >15 years of age now make up more than twenty percent of reported cases. This increase is likely due to several factors, including waning protection from childhood vaccination and natural infection, an increased appreciation for disease in adolescents and adults, and the improved ability of clinicians to diagnose pertussis recognition through the use of serologic methods.

Healthcare workers (HCWs) are at increased risk for acquiring pertussis infection due to regular contact with infected patients and waning protection from childhood vaccination or from natural pertussis infection. Healthcare-associated outbreaks of pertussis have also been increasingly recognized and have been reported from a diverse range of healthcare facilities. Such outbreaks are often due to under-recognition of pertussis with subsequent failure to isolate suspected cases, waning immunity from childhood vaccination or disease, and the increasing incidence of pertussis infection in adults and adolescents. Infected HCWs can then serve as vectors of infection to other susceptible contacts including patients, other employees, and even their own children.

Vaccination is an effective tool for the prevention of pertussis. In 2005, two tetanus toxoid, reduced diphtheria toxoid, and reduced antigen quantity acellular pertussis vaccines (Tdap) were licensed for use in adolescents and adults. In view of the increasingly recognized problem of healthcare-associated and transmitted pertussis infection, the Centers for Disease Control and Prevention's (CDC) Advisory Committee on Immunization Practices (ACIP) targeted HCWs as a priority group for pertussis vaccination in 2006, primarily to reduce the risk of spread of pertussis within health care institutions.

Until the licensure of Tdap, the only method to reduce transmission of pertussis after healthcare-associated exposure to persons with pertussis was post-exposure prophylaxis (PEP) with antibiotics and employee furlough. Close contacts exposed to a pertussis-infected patient or staff member are routinely treated with macrolide therapy (erythromycin or azithromycin), and exposed HCWs who develop a cough-illness are restricted from work for 5 days while on antibiotic therapy. PEP is believed to prevent symptomatic infection in the exposed person if administered within 21 days of cough onset. Traditionally, decisions regarding PEP for exposed HCWs involve detailed assessments of the degree of patient contact, the risk for development of severe or complicated pertussis, and regular evaluation and follow-up for the occurrence of symptoms. These are often time-consuming efforts that are usually the responsibility of infection control or occupational health personnel. With the licensure of Tdap and with the recommended vaccination of HCWs, it is now hoped that vaccination will eliminate the need to provide antibiotic PEP, particularly in recently-vaccinated HCWs. However, this has not been confirmed with a randomized clinical trial, and, therefore, no definitive formal recommendation can be made regarding modifications of PEP in vaccinated HCWs. Two potential strategies exist for the management of vaccinated HCWs following an exposure to a person with pertussis: a) provision of universal antibiotic therapy or b) careful daily observation of vaccinated HCWs for the development of symptoms without antibiotic prescription. A comparison of these two strategies will be the focus of this study.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 - 64 years
* HCW (defined as any healthcare provider with direct patient care duties) who works at VCH (may be primary or secondary place of employment)
* Willing to sign informed consent and authorization for release of information to the Occupational Health Clinic (OHC) at Vanderbilt University
* Planning to work at VCH for at least one year after enrollment or until anticipated study termination, whichever comes first
* Willing to cooperate with disease and microbiologic surveillance

Exclusion Criteria:

* Prior receipt of an acellular pertussis vaccine within 5 years prior to enrollment, unless received since Tdap licensure on June 13, 2005
* History of tetanus booster in the 2 years prior to enrollment (excluding Tdap)
* History of allergic or adverse reaction to diphtheria, tetanus, or pertussis vaccines
* Current pregnancy or attempting to become pregnant in the month after enrollment
* Any contraindication to receipt of pertussis vaccine as listed in the ADACEL package insert
* Febrile illness with temperature greater than 38 degrees C in the previous 72 hours (defer enrollment)
* Persons receiving erythromycin, azithromycin, or related antibiotic for prolonged use
* Persons allergic to both macrolide antibiotics (e.g., azithromycin, clarithromycin, erythromycin) and sulfa antibiotics
* Any condition which, in the opinion of the investigators, may interfere with the evaluation of the study objectives

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1102 (Actual)
Dates: Start 2007-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Talbot, MD MPH, Principal Investigator — Vanderbilt University School of Medicine
Locations (1):
- Monroe Carell Jr. Children's Hospital at Vanderbilt, Vanderbilt University Medical Center,, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Goins WP, Edwards KM, Vnencak-Jones CL, Rock MT, Swift M, Thayer V, Schaffner W, Talbot TR. A comparison of 2 strategies to prevent infection following pertussis exposure in vaccinated healthcare personnel. Clin Infect Dis. 2012 Apr;54(7):938-45. doi: 10.1093/cid/cir973. Epub 2012 Jan 11. PMID 22238169

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between May 2007 and October 2009, all HCWs working at a 206-bed, tertiary care pediatric acute care hospital were recruited for enrollment. Inclusion criteria were age 18 - 64 years; self-report of direct patient contact; planning to work at least one year from enrollment; and willing to cooperate with surveillance.
Pre-assignment Details: Subjects were excluded from randomization if they had a previous pertussis exposure within the past 4 weeks; fever, cough, sore throat, or rhinorrhea; received PEP outside of the study; had been vaccinated with Tdap <7 days prior to the exposure; or were recognized as exposed ≥5 days after identification of the infected patient.
Groups:
- No PEP: Enrolled subjects involved in a pertussis exposure who received no antibiotic post-exposure prophylaxis as per standard recommendations (i.e. azithromycin 500mg x 1 day followed by 250mg Q day for on days 2-5 or trimethoprm sulfamethoxasole DS BID for 14 days)
- Antibiotic PEP: Enrolled subjects involved in a pertussis exposure who received post-exposure prophylaxis as per standard recommendations (i.e. azithromycin 500mg x 1 day followed by 250mg Q day for on days 2-5 or trimethoprm sulfamethoxasole DS BID for 14 days)
Period: Overall Study
Arm/Group | No PEP | Antibiotic PEP
Started | 44 | 42
Completed | 44 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No PEP | Antibiotic PEP | Total
Number analyzed (Participants) | 44 | 42 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 42 | 86
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32 (2) | 27 (2) | 29 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 29 | 55
  Male | 18 | 13 | 31
Region of Enrollment [Number; unit: participants]
  United States | 44 | 42 | 86

OUTCOME MEASURES:

1. Primary Outcome: Evidence of Pertussis Infection in Each PEP Arm, Defined Using Clinical, Microbiologic, or Serologic Criteria.
Description: Defined as a positive nasopharyngeal culture or PCR for B. pertussis at any time point, a two-fold rise in the anti-PT IgG titer between acute and convalescent sera, or a single acute or convalescent anti-PT IgG titer of ≥94 EU. Post hoc, a modified definition was devised because of concern that the serologic criteria used in the primary definition might actually represent acquisition of pertussis infection prior to the intervention. The modified definition of pertussis excluded an acute anti-PT IgG titer of ≥94 EU and an acute nasopharyngeal swab that was positive for B. pertussis by PCR.
Time Frame: In the 21 days following exposure identification
Measure: Number; unit: participants
Arm/Group | No PEP | Antibiotic PEP
Number analyzed (Participants) | 44 | 42
participants | 6 | 1

ADVERSE EVENTS:
Arm/Group | No PEP | Antibiotic PEP
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/42
Other Adverse Events (participants affected / at risk) | 0/44 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No